CLINICAL TRIAL: NCT05926700
Title: Efficacy and Safety of Cadonilimab Combined With Anlotinibin in the Treatment of Advanced or Metastatic Soft Tissue Sarcoma With Previous First-Line Standard Treatment Failure.
Brief Title: Efficacy and Safety of Cadonilimab Plus Anlotinib in Advanced STS That Failed the Previous First-line Standard Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0454
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): The subject will be treated with Candonilimab + anlotinib every 21 days as a treatment cycle: Candonilimab 10mg/kg, D1 administration; Anlotinib 12mg/ day was taken orally for 2 weeks and stopped for a week. Until the subject has disease progression, intolerable toxicity, and the investigator's decision, the subject withdraws informed consent, death or other reasons specified in the protocol.
  Interventions: Drug: Candonilimab

INTERVENTIONS:
Drug: Candonilimab — The patients were treated with Candonilimab + anlotinib, with Cadonilimab 10mg/kg, D1 administration; Anlotinib 12mg/ day was orally administered for 2 weeks and stopped for a week, with 21 days as a course of treatment.

SUMMARY:
Objective to evaluate the efficacy and safety of candonilimab combined with anlotinib in the treatment of progressive or metastatic soft tissue sarcoma that failed previous first-line standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 70 years (including 18 and 70).
2. Voluntarily sign written informed consent.
3. Advanced or unresectable soft tissue sarcomas confirmed by pathology mainly include liposarcoma, leiomyosarcoma, synovial sarcoma, undifferentiated pleomorphic sarcoma / malignant fibrous histiocytoma, fibrosarcoma, pleomorphic rhabdomyosarcoma, acinar soft tissue sarcoma, clear cell sarcoma, angiosarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumor, undifferentiated sarcoma, sarcoma after radiotherapy, etc.
4. Patients who have used at least one chemotherapy regimen (including anthracyclines) in the past (except for acinar soft tissue sarcoma and clear cell sarcoma) and are evaluated as disease progression according to the efficacy evaluation criteria of solid tumors within 6 months.
5. According to RECIST 1.1, there was at least one measurable tumor lesion.
6. ECoG score 0 or 1.
7. The expected survival was ≥ 3 months.
8. The main organs function well:

   a) Hematology (no blood components and cell growth factors were used to support treatment within 7 days before starting the study treatment):

   i. The absolute value of neutrophils ANC ≥ 1.5 × 109/l (1500/mm3).

   Ii Platelet count ≥ 100 × 109/l (100000/mm3).

   III. hemoglobin ≥ 90 g/l.

   b) Kidney:

   i. Creatinine clearance * (CrCl) calculated value ≥ 50 ml/min.

   *The Cockcroft Gault formula will be used to calculate CrCl (Cockcroft Gault formula)

   CrCl (ml/min) = [(140 - age) × Weight (kg) × F] / (SCR (mg/dl) × 72)

   Among them, f=1 for men and f=0.85 for women; SCR = serum creatinine.

   Ii Urine protein < 2+ or 24-hour (H) urine protein quantification <1.0 G.

   c) Liver:

   i. Total serum bilirubin (TBIL) ≤ 1.5 × ULN.

   II. AST and alt ≤ 2.5 × ULN.

   III. for subjects with liver metastasis, serum total bilirubin (TBIL) ≤ 3 × ULN; ALT and AST ≤ 5 × ULN;

   d) Coagulation function:

   i. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
9. Female subjects with fertility must have a serum pregnancy test within 3 days before the first medication and the result is negative. If a female issue with fertility has sex with a male partner who has not been sterilized, the subject must take an acceptable contraceptive method since the screening, and must agree to continue using the contraceptive method within 6 months after the last administration of the study drug; Whether to stop contraception after this time point should be discussed with the investigator.
10. The subject is willing and able to comply with the visit, treatment plan, laboratory test, and other study requirements as stipulated in the schedule.

Exclusion Criteria:

1. Participated in the treatment of experimental drugs or used experimental devices within 4 weeks before the first administration of candonilimab.
2. Had other active malignancies within 3 years before enrollment. Except for locally curable malignant tumors (manifested as cured), such as basal or cutaneous squamous cell carcinoma, superficial bladder cancer, endometrial, cervical or breast cancer in situ.
3. Another clinical study is enrolled at the same time, unless it is an observational (non interventional) clinical study or the follow-up period of an interventional study (defined as the time from the first medication to the last medication of the previous clinical study is more than 4 weeks or the five half lives of the study drug are more than 5, whichever is the longest).
4. Active autoimmune diseases requiring systemic treatment within two years before the start of study treatment, or autoimmune diseases that may recur or are planned to be treated according to the judgment of the investigator; The following exceptions: skin diseases that do not need systematic treatment (such as vitiligo, alopecia, psoriasis or eczema); Hypothyroidism caused by autoimmune thyroiditis only requires a stable dose of hormone replacement therapy; Well controlled type I diabetes; Subjects whose asthma in childhood has been completely relieved and who do not need any intervention after adulthood; The investigator judged that the disease would not recur without external triggers.
5. Inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea) with active or requiring clinical treatment.
6. The subject required systemic treatment with corticosteroids (>10mg daily prednisone equivalent) or other immunosuppressive drugs within 14 days after taking the study drug. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal gland replacement doses of >10mg daily prednisone equivalent were allowed. Subjects were allowed to use topical, ocular, intra-articular, intranasal, and inhaled corticosteroids (with minimal systemic absorption). Physiological alternative doses of systemic corticosteroids are allowed, even if >10 mg / day of prednisone equivalent. Short term use of corticosteroids is allowed to prevent (such as contrast allergy) or treat non autoimmune diseases (such as delayed type hypersensitivity caused by contact allergens).
7. He has previously received immune checkpoint inhibitors (such as anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.), immune checkpoint agonists (such as antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.), immune cell therapy and other treatments targeting tumor immune mechanism.
8. The best swelling evaluation result of patients who had received previous treatment with anlotinib was PD, or SD ≤ 12 weeks.
9. History of a known positive test for human immunodeficiency virus or known acquired immune deficiency syndrome.
10. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
11. Known presence or history of interstitial lung disease.
12. Necrotic lesions were found within 4 weeks before the subjects were enrolled, and the investigator judged that there was a risk of major bleeding.
13. Serious infections occurred within 4 weeks before the first administration, including but not limited to complications requiring hospitalization, sepsis or severe pneumonia.
14. Known to have active pulmonary tuberculosis (TB). Subjects suspected of active TB should be examined by chest X-ray, sputum and excluded by clinical symptoms and signs.
15. Untreated patients with chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA > 1000iu/ml, and patients with active hepatitis C should be excluded. Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV dna<1000iu/ml), and cured hepatitis C patients can be enrolled. For HCV AB positive subjects, they are eligible to participate in the study only if HCV RNA test results are negative.
16. Received the last radiotherapy or anti-tumor treatment (chemotherapy, targeted therapy, Chinese herbal medicine used to control tumor disease or tumor embolization, etc.) within 4 weeks before the first administration of candonilimab.
17. Major surgical procedures were performed within 30 days before the first dose of candonilimab or had not yet fully recovered from previous surgery. Local surgery (such as systemic port placement, core needle biopsy, and prostate biopsy) was allowed, provided that the surgery was completed at least 24 hours before the first administration of the study treatment drug.
18. Meningeal metastasis, spinal cord compression, leptomeningeal disease, or active brain metastasis are known. However, subjects who meet the following requirements and have measurable lesions outside the central nervous system are allowed to be enrolled: 1) they have not been treated before and are currently asymptomatic (such as no neurological dysfunction, epilepsy or other typical symptoms and signs of central nervous system metastasis; no glucocorticoid treatment is required); 2) After treatment, the patient was asymptomatic, and the imaging was stable for at least 4 weeks before the start of study treatment (if there were no new or expanded brain metastases), and the treatment of systemic glucocorticoids and anticonvulsants had been stopped for at least 2 weeks.
19. According to the judgment of the investigator, subjects with pleural effusion, pericardial effusion or ascites that cannot be stably controlled by repeated drainage or other methods.
20. Uncontrolled concurrent diseases, including symptomatic congestive heart failure (grade 3 or 4 according to the New York Heart Association functional classification), uncontrolled hypertension, unstable angina, poorly controlled arrhythmia, evidence of acute or ongoing myocardial ischemia, severe active peptic ulcer disease or gastritis, Or mental illness / social condition that will restrict subjects' compliance with research requirements or affect subjects' ability to provide written informed consent. Any arterial thromboembolic event occurred within 6 months before enrollment, including myocardial infarction, cerebrovascular accident or transient ischemic attack, with a history of deep vein thrombosis, pulmonary embolism or any other serious thromboembolism.
21. the toxicity of previous anti-tumor treatment was not relieved, which was defined as the toxicity did not return to grade 0 or 1 of NCI CTCAE version 5.0, or the level specified in the inclusion / exclusion criteria, except for hair loss. Subjects who have irreversible toxicity and are not expected to aggravate after the administration of study drugs (such as hearing loss) may be included in the study after consultation with the medical inspector. Subjects with long-term toxicity caused by radiotherapy who cannot recover according to the judgment of the investigator may be included in the study after consultation with the medical inspector.
22. received a live vaccine within 30 days before the first dose of candonilimab or planned to receive a live vaccine during the study period.
23. known history of severe hypersensitivity to other monoclonal antibodies.
24. are known to be allergic to any of the components of the candonilimab formulation.
25. pregnant or lactating women.
26. any condition that the investigator believes may lead to the risk of receiving study drug treatment, or will interfere with the evaluation of study drug or the safety of subjects or the analysis of study results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | through study completion，an average of 1 year
  The proportion of patients whose tumor volume reduced by 30% and could maintain for more than 4 weeks, that is, the sum of the proportion of complete remission (CR) and partial remission (PR)

SECONDARY OUTCOMES:
disease control rate （DCR) | through study completion，an average of 1 year
  The percentage of disease remission (including complete remission and partial remission, pr+cr) and stable disease (SD) in the number of evaluable cases after treatment
Duration of Response(DOR) | through study completion，an average of 1 year
  Remission duration refers to the time from the first CR or PR to disease progression.
time-to-response (TTR) | through study completion，an average of 1 year
  It refers to the overall time from the time of tumor occurrence to the patient's death
Progression-Free-Survival （PFS） | through study completion，an average of 1 year
  Time from randomization to disease progression
Overall survival （OS） | through study completion，an average of 1 year
  The overall survival time of tumor patients
Adverse events | through study completion，an average of 1 year
  The incidence and severity of adverse events (AES) and clinically significant abnormal laboratory test results.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Dong, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China